CLINICAL TRIAL: NCT04451356
Title: The Complex Evaluation of the Cardiovascular Risk in the Kidney Transplant Patients
Brief Title: Romanian Kidney Transplant Cardiovascular Risk Registry
Acronym: ROKET-CV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Dimitrie Siriopol, Associate Professor, Grigore T. Popa University of Medicine and Pharmacy
Other Study IDs: UMF
Record Dates: First submitted 2019-10-08; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Kidney Transplant; Complications; Cardiovascular Diseases
Keywords: Kidney Transplant; Bioimpedance Spectroscopy; Arterial stiffness
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Bioimpedance Spectroscopy — This analysis will be performed at baseline using the portable whole-body multifrequency bioimpedance analysis device (BCM®Body Composition Monitor - Fresenius Medical Care D GmbH). The technique involves attaching electrodes to the patient's forearm and ipsilateral ankle, with the patient in a supine position. The BCM® measures the body resistance and reactance to electrical currents of 50 discrete frequencies, ranging between 5 and 1000 kHz. Based on a fluid model using these resistances, the extracellular water (ECW), the intracellular water (ICW) and the total body water (TBW) are calculated. These volumes are then used to determine the amount of fluid overload. All calculations are automatically performed by the software of the BCM® device. In addition, this analysis will provide the LTI and FTI for the included patients.
Device: Arterial Stiffness — Arterial stiffness assessment will be performed by applanation tonometry (SphygmoCorTM; PWV Inc., Westmead, Sydney, Australia) with the patient being recumbent, 10 minutes before the measures were done. The carotid and femoral pulse will be acquired by applanation tonometry sequentially, allowing a single operator to acquire the measurement. The transit time from the R-wave of the simultaneously acquired electrocardiogram to the foot of the carotid and femoral pulse is measured. The difference acquired electrocardiogram to the foot of the carotid and femoral pulse is measured. The difference between these 2 transit times is divided by distances measured from the body surface to estimate the arterial path length in order to calculate carotid-femoral PWV.
Diagnostic Test: Echocardiography — Echocardiographic evaluations will be made in each patient at baseline. All echocardiographic measurements will be carried out according to the recommendations of the American Society of Echocardiography by an observer unaware of the lung ultrasound and bioimpedance results. Echocardiographic evaluation will provide information about cardiac anatomy (e.g. volumes, geometry, mass) and function (e.g. left ventricular function and wall motion, valvular function, right ventricular function, pulmonary artery pressure, pericardium).
Diagnostic Test: Lung ultrasonography — Examinations will be performed in the supine position. Scanning of the anterior and lateral chest will be performed on both sides of the chest, from the second to the fourth (on the right side to the fifth) intercostal spaces, at parasternal to mid-axillary lines. B-lines will be recorded in each intercostal space and were defined as a hyperechoic, coherent US bundle at narrow basis going from the transducer to the limit of the screen. B-lines starting from the pleural line can be either localized or scattered to the whole lung and be present as isolated or multiple artifacts. The sum of B-lines produces a score reflecting the extent of lung water accumulation (0 being no detectable B-line).

SUMMARY:
Kidney transplantation (KT) represents the best treatment for patients with end-stage kidney disease, being associated with improved outcomes and reduced mortality. Although the survival benefit with KT is mostly attributable to reduction in cardiovascular (CV) disease, KT recipients continue to remain at higher risk for CV-related morbidity and mortality when compared with the general population. Additionally, CV events represent the leading cause of death in KT recipients with a functioning allograft. KT recipients have high rates of hospitalization for myocardial infarction, congestive heart failure, dysrhythmias, stroke, malignant hypertension, and cardiac arrest. Significant amounts of research have been aimed at reducing event rates, primarily aimed at understanding prevalent risk factors, defining outcomes, and application of guideline-based care.

The post-KT milieu represents the confluence of several traditional and nontraditional CV risk factors contributing to the significant CV risk in this population. CV disease remains an understudied and undertreated source of morbidity and mortality in KT patients. Patients with chronic kidney disease (CKD) are generally excluded from major cardiovascular outcome trials, and this phenomenon of aversion to including patients with CKD in CV trials and providing appropriate goal-directed medical and interventional therapies (renalism) extends into KT .

The main aim of this study is to evaluate holistically the CV risk in a KT population. The investigators will compare bioimpedance spectroscopy derived fluid status parameters (overhydration, total body water, extracellular water and intracellular water) with clinical evaluation, lung ultrasonography, pulse wave velocity, different biomarkers, and echocardiographic characteristics and also to determine the impact of these parameters on renal and CV outcomes in the same population.

DETAILED DESCRIPTION:
• Patients:

The inclusion criteria are:

1. age>18 years;
2. KT recipient.

The exclusion criteria are:

1. metallic joint prostheses, cardiac stent or pacemakers, decompensated cirrhosis, pregnancy and limb amputations (due to bioimpedance technique limitations);
2. no prior diagnosis of pulmonary fibrosis, pneumectomy or massive pleural effusion (due to lung ultrasonography limitations);
3. active systemic infections (due to difficulties in the interpretation of nespecific inflammation biomarkers in this type of patients);
4. absence of congenital heart disease;
5. eGFR below 30 ml/min/1.73m2;
6. KT vintage of at least 6 months.

   * Methods:

All patients will have a complete clinical and paraclinical evaluation:

* Personal data (age, sex, height);
* Cardiovascular risk factors (smoking, weight, body mass index);
* Medication (including immunosupression);
* Kidney transplantation data (date of transplantation, type - living or cadaveric donor, missmatch number, type of induction therapy);
* Dialysis vintage (before KT)
* Comorbidities (diabetes, hypertension, stroke, coronary artery disease, etc);
* Physical examination (blood pressure, crackles, pedal edema etc);
* Renal function evaluation (serum urea and creatinine, serum electrolytes - K, Na, Cl)
* Nutrition status evaluation: serum protein, cholesterol, triglycerides;
* Inflammation evaluation: CRP;
* Serum glucose and uric acid;
* Hemoleucogram;
* Electrocardiogram.

Bioimpedance spectroscopy analysis This analysis will be performed at baseline using the portable whole-body multifrequency bioimpedance analysis device (BCM®Body Composition Monitor - Fresenius Medical Care D GmbH). The technique involves attaching electrodes to the patient's forearm and ipsilateral ankle, with the patient in a supine position. The BCM® measures the body resistance and reactance to electrical currents of 50 discrete frequencies, ranging between 5 and 1000 kHz. Based on a fluid model using these resistances, the extracellular water (ECW), the intracellular water (ICW) and the total body water (TBW) are calculated. These volumes are then used to determine the amount of fluid overload. All calculations are automatically performed by the software of the BCM® device. Absolute fluid overload (AFO) is is defined as the difference between the expected patient's ECW under normal physiological conditions and the actual ECW, whereas the relative fluid overload (RFO) is defined as the absolute fluid overload AFO to ECW ratio. Normohydration is defined when AFO is between the 10th and the 90th percentile for healthy, age- and gender-matched individuals from the reference population, i.e. between -1.1 to +1.1 L, while volumes below and above this range defining underhydration and overhydration, respectively. In addition, this analysis will provide the LTI and FTI for the included patients.

Echocardiography Echocardiographic evaluations will be made in each patient at baseline. All echocardiographic measurements will be carried out according to the recommendations of the American Society of Echocardiography by an observer unaware of the lung ultrasound and bioimpedance results. Echocardiographic evaluation will provide information about cardiac anatomy (e.g. volumes, geometry, mass) and function (e.g. left ventricular function and wall motion, valvular function, right ventricular function, pulmonary artery pressure, pericardium).

Lung ultrasonography Examinations will be performed in the supine position. Scanning of the anterior and lateral chest will be performed on both sides of the chest, from the second to the fourth (on the right side to the fifth) intercostal spaces, at parasternal to mid-axillary lines. B-lines will be recorded in each intercostal space and were defined as a hyperechoic, coherent US bundle at narrow basis going from the transducer to the limit of the screen. B-lines starting from the pleural line can be either localized or scattered to the whole lung and be present as isolated or multiple artifacts. The sum of B-lines produces a score reflecting the extent of lung water accumulation (0 being no detectable B-line).

Arterial stiffness Arterial stiffness assessment will be performed by applanation tonometry (SphygmoCorTM; PWV Inc., Westmead, Sydney, Australia) with the patient being recumbent, 10 minutes before the measures were done. The carotid and femoral pulse will be acquired by applanation tonometry sequentially, allowing a single operator to acquire the measurement. The transit time from the R-wave of the simultaneously acquired electrocardiogram to the foot of the carotid and femoral pulse is measured. The difference acquired electrocardiogram to the foot of the carotid and femoral pulse is measured. The difference between these 2 transit times is divided by distances measured from the body surface to estimate the arterial path length in order to calculate carotid-femoral PWV. The SphygmoCor PWV has been established in the literature as a reference for comparison due to the wealth of population data and healthy population refence values. The investigators will determine two PWVs for every patient and use the media for the statistical analysis. If the difference between these two measurements will be higher than 0.5 m/s then another determination will be performed and the median will be used for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. age>18 years;
2. Kidney Transplant Recipient.

Exclusion Criteria:

1. metallic joint prostheses, cardiac stent or pacemakers, decompensated cirrhosis, pregnancy and limb amputations (due to bioimpedance technique limitations);
2. no prior diagnosis of pulmonary fibrosis, pneumectomy or massive pleural effusion (due to lung ultrasonography limitations);
3. active systemic infections (due to difficulties in the interpretation of nespecific inflammation biomarkers in this type of patients);
4. absence of congenital heart disease;
5. eGFR below 30 ml/min/1.73m2;
6. KT vintage of at least 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney Transplant Recipients
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Composite Renal Outcome | 36 months
  Doubling of creatinine or dialysis initiation.
Composite Cardiovascular Outcome | 36 months
  Time to first non-fatal myocardial infarction, non-fatal stroke, hospitalization for heart failure, or cardiovascular death

SECONDARY OUTCOMES:
Chronic kidney disease progression | 36 months
  The impact of baseline characteristics on eGFR (as assessed by the CKD-EPI formula) evolution
Proteinuria progression | 36 months
  The impact of baseline characteristics on proteinuria (as assessed by the urine protein to creatinine ratio) evolution

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Covic, Prof, Study Chair — Grigore T. Popa University of Medicine and Pharmacy, Iasi
Locations (1):
- "Dr. C.I. Parhon" Hospital, Iași, Romania

IPD SHARING:
Plan to Share IPD: Undecided